CLINICAL TRIAL: NCT02642692
Title: Hamstrings X Patellar Tendon for Anterior Cruciate Ligament Reconstruction in Soccer Players - RCT
Brief Title: Hamstrings X Patellar Tendon for ACL Reconstruction in Soccer Players - RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Luiz Gabriel Betoni Guglielmetti, MD, Master, Phd, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16373713.1.0000.5479
Record Dates: First submitted 2015-12-25; First posted 2015-12-30 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL reconstruction; Single bundle; Clinical results; Soccer players
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patellar Tendon Graft (Experimental): Kind of graft that will be used for acl reconstruction
  Interventions: Procedure: Patellar Tendon graft
- Hamstring Graft (Experimental): Kind of graft that will be used for acl reconstruction
  Interventions: Procedure: Hamstring Graft

INTERVENTIONS:
Procedure: Patellar Tendon graft — Acl reconstruction with patellar tendon graft
  Arms: Patellar Tendon Graft
Procedure: Hamstring Graft — Acl reconstruction with hamstring graft
  Arms: Hamstring Graft

SUMMARY:
The purpose of this study is to specifically evaluate outcomes of bone-patellar tendon-bone autograft versus hamstring autograft ACL reconstruction in soccer players.

DETAILED DESCRIPTION:
A number of techniques for ACL reconstruction have been proposed and tested, and most surgeons now prefer autografts with the patellar tendon or semitendinosus tendon. The functional outcome after ACL reconstruction with the patellar or semitendinosus tendon has been a recent area of interest. Soccer is the most popular sport worldwide with more than 260 million active players, and it is hard to say if patellar tendon or semitendinosus grafts have different outcomes.

The purpose of this study was to specifically evaluate outcomes of bone-patellar tendon-bone autograft versus hamstring autograft ACL reconstruction in soccer players. The hypothesis of this study was that hamstring autograft ACL reconstruction would provide no statistically significant differences in patient-reported outcome scores, postoperative level of sports function, and harvest-site morbidity when compared with patellar tendon autograft .The Cincinnati Knee Rating System (CKRS) was chosen as the primary outcome. As secondary outcome, reruptures.

Between march 2016 and march 2017, 60 soccer players will be operated. The investigators consider as soccer players those who play more than 4 times a week. Once included in the study, they will be randomized in two groups: "hamstring group" and "patellar tendon group".

The final clinical evaluation with two years. For both groups, the technique is the same, the fixation of the grafts with metal interference screws. Femoral tunnel will be drilled with outside-in technique. The tibial tunnel with conventional 55 degrees guide.

Both groups of patients will receive the same physical therapy protocol. Data will be evaluated with the SPSS software for Windows (version 13.0).

ELIGIBILITY:
Inclusion Criteria:

* unilateral ACL lesion
* skeletally mature patients with closed physis
* no previous surgery on the affected knee (except for arthroscopic meniscectomy)
* less than 1 year from injury
* no associated ligament injuries (except for the medial collateral ligament grade I and II)
* soccer players.

Exclusion Criteria:

* morbid obesity
* degenerative changes in arthroscopy or image exams
* those who play soccer less than 4 times / week

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Cincinnati Knee Rating System | 2 years
  It is a subjective score

SECONDARY OUTCOMES:
rerupture | 2 years
International Knee Documentantion Committee (IKDC) score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: luiz G guglielmetti, MD, Principal Investigator — Faculdade de Ciencias Medicas da Santa Casa de São Paulo
Locations (1):
- Faculdade de Ciencias Medicas da Santa Casa de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corry IS, Webb JM, Clingeleffer AJ, Pinczewski LA. Arthroscopic reconstruction of the anterior cruciate ligament. A comparison of patellar tendon autograft and four-strand hamstring tendon autograft. Am J Sports Med. 1999 Jul-Aug;27(4):444-54. doi: 10.1177/03635465990270040701. PMID 10424213
- [Background] Aglietti P, Buzzi R, Zaccherotti G, De Biase P. Patellar tendon versus doubled semitendinosus and gracilis tendons for anterior cruciate ligament reconstruction. Am J Sports Med. 1994 Mar-Apr;22(2):211-7; discussion 217-8. doi: 10.1177/036354659402200210. PMID 8198189
- [Background] Carter TR, Edinger S. Isokinetic evaluation of anterior cruciate ligament reconstruction: hamstring versus patellar tendon. Arthroscopy. 1999 Mar;15(2):169-72. doi: 10.1053/ar.1999.v15.0150161. PMID 10210074
- [Background] Mascarenhas R, Tranovich MJ, Kropf EJ, Fu FH, Harner CD. Bone-patellar tendon-bone autograft versus hamstring autograft anterior cruciate ligament reconstruction in the young athlete: a retrospective matched analysis with 2-10 year follow-up. Knee Surg Sports Traumatol Arthrosc. 2012 Aug;20(8):1520-7. doi: 10.1007/s00167-011-1735-2. Epub 2011 Nov 3. PMID 22048746
- [Background] Walden M, Hagglund M, Werner J, Ekstrand J. The epidemiology of anterior cruciate ligament injury in football (soccer): a review of the literature from a gender-related perspective. Knee Surg Sports Traumatol Arthrosc. 2011 Jan;19(1):3-10. doi: 10.1007/s00167-010-1172-7. Epub 2010 Jun 9. PMID 20532868
- [Background] Fink C, Hoser C, Benedetto KP, Judmaier W. [(Neuro)muscular changes in the knee stabilizing muscles after rupture of the anterior cruciate ligament]. Sportverletz Sportschaden. 1994 Mar;8(1):25-30. doi: 10.1055/s-2007-993449. German. PMID 8197541
- [Derived] Guglielmetti LGB, Salas VER, Jorge PB, Severino FR, Duarte A, de Oliveira VM, Cury RPL. Prospective and Randomized Clinical Evaluation of Hamstring Versus Patellar Tendon Autograft for Anterior Cruciate Ligament Reconstruction in Soccer Players. Orthop J Sports Med. 2021 Sep 24;9(9):23259671211028168. doi: 10.1177/23259671211028168. eCollection 2021 Sep. PMID 34604426